CLINICAL TRIAL: NCT05025293
Title: Zoledronate Early to Hip Fracture Patients - Safe and Effective? A Double-blinded Randomized Controlled Treatment Strategy Trial on Zoledronate in Hip Fracture Patients
Brief Title: Zoledronate Early to Hip Fracture Patients - Safe and Effective?
Acronym: ZEBRA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lene Bergendal Solberg (Other)
Collaborators: Vestre Viken Hospital Trust (Other); Roche Diagnostics GmbH (Industry); Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor-Investigator, Lene Bergendal Solberg, Principal Investigator, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2018/2234; 2020-000638-17 (EudraCT Number)
Record Dates: First submitted 2021-08-18; First posted 2021-08-27 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Hip Fractures; Osteoporosis
Keywords: hip fractures; zoledronic acid; bone turnover markers; delirium; early rehabilitation; bone mineral density
MeSH Terms: conditions — Hip Fractures; Osteoporosis; Delirium | interventions — Zoledronic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled non-inferiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patients are randomized by an electronic system (Viedoc). The randomization is masked for the investigator, the care providers, the participants and the outcomes assessor. Only un-blinded authorized study personnel who prepare the study medicine will see the allocation. The study medicine will be kept in a locked box. Blinded authorized personnel will give the study medication to the patients. The infusions will be covered by a locked box not allowing the patients or others to know the type of infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZOLearly (Experimental): Within 3 days after hip fracture surgery: A single dose of 100 ml containing 5mg zoledronate (Aclasta) will be administered intravenously.
  The ZOLearly group will have no further infusions during the study period.
  Interventions: Drug: Zoledronic Acid 5Mg/Bag 100Ml Inj
- ZOLlate (Placebo Comparator): Within 3 days after hip fracture surgery: A single dose of 100 ml containing 100ml NaCl 9mg/ml (placebo) will be administered intravenously.
  3 months after hip fracture surgery (at the out-patient clinic): A single dose of 100 ml containing 5mg zoledronate (Aclasta) will administered intravenously.
  Interventions: Drug: Zoledronic Acid 5Mg/Bag 100Ml Inj; Drug: sodium chloride

INTERVENTIONS:
Drug: Zoledronic Acid 5Mg/Bag 100Ml Inj — 100ml Zoledronic acid (5mg/100ml) administered intravenously
  Other Names: Zoledronate; Aclasta
Drug: sodium chloride — 100ml NaCl 9mg/ml administered intravenously
  Other Names: NaCl
  Arms: ZOLlate

SUMMARY:
To prevent hip fracture patients for having another fracture, secondary fracture preventing medication should be given as soon as possible. Zoledronate is the most efficient bisphosphonate and is given as an intravenous infusion once yearly. However, the appropriate time to initiate zoledronate treatment after a hip fracture has not yet been established. To clarify the optimal timing of zoledronate to hip fracture patients we have designed a double-blinded, placebo-controlled randomized non-inferiority trial to compare if zoledronate administered early (within 5 days) after hip fracture surgery is as good as zoledronate given late (3 months) after hip fracture surgery.

DETAILED DESCRIPTION:
Hip fracture patients have the highest risk for recurrent hip or other osteoporotic fractures. We have efficient fracture preventing medication easily available, but few patients receive them. We therefore need to create simple systems to ensure that these frail patients with the highest risk for a new fracture are offered proper treatment early and any delay in treatment should be avoided. Zoledronate is the most efficient bisphosphonate and the drug of choice for hip fracture patients due to the results from the Horizon recurrent fracture trial. It is given as an intravenous infusion once yearly. However, the appropriate time to initiate zoledronate treatment after a hip fracture has not yet been established. The summary of product characteristics (SmPC) for Aclasta (zoledronate) in Norway says that Aclasta should not be administered within the first 2 weeks after the hip fracture, however there have been a practice over years in Norway to give zoledronate to the hip fracture patients during their stay in hospital for fracture treatment. There are logistical and practical advantages of giving zoledronate while the patient is still in hospital for her fracture. It has, however, been questioned whether the effect of zoledronate given within the first 2 weeks postoperatively really is fracture preventing. The results from the post hoc analysis from the Horizon recurrent fracture trial by Eriksen and co-workers in 2009, suggested that given zoledronate within 2-weeks after hip fracture surgery may be a little less fracture preventing. The results from this analysis can be due to the low number of study subjects as well as frailty in the study population causing the large variations. On the other hand, the lack of effect in the within 2-week group may be due to the affinity for zoledronate to bone mineral and the accumulation of zoledronate in the fracture callus during bone repair with less being incorporated in the rest of the skeleton.

To clarify the optimal timing of zoledronate to hip fracture patients we wanted to compare if zoledronate administered early (within 5 days) after hip fracture surgery, while the patients is still in hospital, is as good as zoledronate given late (3 months) after hip fracture surgery.

To test our hypothesis we designed a non-inferiority randomized trial using the bone turnover marker N-terminal propeptide of type I procollagen (P1NP) as the primary endpoint. PINP has in recent years been widely used as a marker to follow the effect of anti-resorptive therapy as it is more robust than the other well studied bone marker; cross-linked C-telopeptide of type I collagen (CTX). P1NP and CTX are recommended as reference markers for bone turnover by the International Osteoporosis Foundation (IOF). Anti-resorptive agents as bisphosphonates influence bone remodeling by decreasing bone resorption (amino-bisphosphonates kills osteoclasts) and thereby also reducing bone formation. This affects the bone turnover markers: Both P1NP and CTX drops in value in a consistent manner reflecting the level of bone suppression and has shown to correlate with the level of bone mineral density and the subsequent fracture risk. P1NP and CTX are therefore well suited to monitor the effect of anti-resorptive therapy as they reflect the bone turnover status in the entire skeleton. It is likely to believe that if zoledronate given early after fracture is accumulated in the fracture callus and too little is incorporated in the entire skeleton, the result will be just a local decrease in bone resorption (only in the fracture callus). This will not to the same extent as a decrease in bone resorption from the entire skeleton, be reflected by the bone turnover markers P1NP and CTX and the fall in these markers will be less than if we give zoledronate after the fracture has healed (after 6-12 weeks).

Eligible patients that meets the study requirements and with an informed consent will be stratified on type of operation (arthroplasty versus internal fixation) and on hospital before randomization 1:1 to either zoledronate early (ZOLearly: zoledronate given within 5 days after hip fracture surgery) or zoledronate late (ZOLlate: zoledronate given 3 months after hip fracture surgery). The patients will be followed for 15 months with study visits at 3 months post fracture and at 6 and 12 months post treatment with zoledronate. The study is double-blinded the first 3 months to be able to test for the "soft" secondary endpoints; delirium and rehabilitation. Approximately 300 patients will be recruited. Estimated recruitment time is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Low energy hip fracture
* Surgery within 72 hours
* >50 years old norwegian
* Women age 50-60 must be postmenopausal or not pregnant
* Acceptable kidney function (estimated GFR >=35) and calcium levels
* Fit to complete the follow-up judged by the recruiting physician
* Signed informed consent by the patient or the next of kin

Exclusion Criteria:

* Metal in the opposite hip
* Anti-osteoporosis treatment with bisphosphonates, denosumab, teriparatide, abaloparatide or romosozumab within the last 10 years
* Glucocorticoid therapy
* Too sick to receive treatment with zoledronate judged by the recruiting or treating physician
* Any other contraindication listed on the SmPC of the IMP(s) including pregnancy
* Participating in another trial that might affect the current study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Difference between the two groups (ZOLearly vs ZOLlate) in proportion of patients having P1NP>35µg/L 12 months after treatment with zoledronate | 12 months after treatment with zoledronate
  Measured by the bone turnover marker N-terminal propeptide of type 1 procollagen (P1NP) (µg/ml) in blood samples

SECONDARY OUTCOMES:
Grade of early mobilization | 1-30 days
  Measured by Cumulated Ambulation Score (CAS) in hospital and at discharge from hospital. The score range from 0 to 6, where 6 is the best. The patient is scored daily during the stay in hospital.
Delirium assessment | 1-30 days
  Number of patients with delirium assessed by 4 "A" test (4AT) in hospital
Difference between the two groups in proportion of patients having CTX>0.28µg/L 12 months after treatment with zoledronate | 12 months after treatment with zoledronate
  Measured by the bone turnover marker C-telopeptide of type 1 collagen (CTX) (µg/ml) in blood samples
Change in bone mineral density (BMD) | 12 months after treatment with zoledronate
  Measured by dual-energy x-ray absorbtiometry (DXA) in g/cm2 right after hip fracture surgery and after 12 months with zoledronate treatment
Grade of mobilization and rehabilitation | 3 months after fracture surgery
  Measured by Time-up-and-go (TUG) test
Fever (T> 38'C) during hospital stay for fracture surgery | 1-30 days
  Temperature measured in 'C in each patient
Use of antibiotics during hospital stay for fracture surgery | 1-30 days
  Measure duration of antibiotic treatment in each patient
Hospital stay after hip fracture surgery | 1-30 days
  Measure time from admission to discharge from hospital and time from hip fracture surgery to discharge from hospital
Time to readmission to hospital (any department) after first discharge | 15 months
  Measure time to first readmission for each patient
Number of readmissions to hospital (any department) after first discharge | 15 months
  Measure number of readmissions for each patient
Time to new fracture | 15 months
  Measure time to first new fracture after the index fracture for each patient
Total number of new fractures | 15 months
  Measure total number of new fractures
Deaths | 15 months
  Measure total number of deaths

OTHER OUTCOMES:
Health-related quality of life | 12 months after treatment with zoledronate
  Measured by EQ-5D-5L
Time to fracture healing for the patients with osteosynthesis | 3 months after fracture treatment
  Examined by x-rays and TUG test

CONTACTS AND LOCATIONS:
Overall Officials: Solberg B Lene, PhD MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway